CLINICAL TRIAL: NCT00618176
Title: Three Generic Nevirapine-Based Antiretroviral Treatments in Chinese Patients:Multicentric Observation Cohort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Taisheng Li, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004BA719A10; 2004BA719A10
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; adverse effects; Treatment Outcome; Drug Resistance, Viral; treatment naïve
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Stavudine; Lamivudine; Nevirapine

ARMS (3):
- B (Experimental)
  Interventions: Drug: Stavudine (d4T), Lamivudine (3TC), Nevirapine (NVP)
- A (Experimental)
  Interventions: Drug: Zidovudine (AZT)+ Didanosine (ddI)+ Nevirapine (NVP)
- C (Experimental)
  Interventions: Drug: Zidovudine (AZT), Lamivudine (3TC), Nevirapine (NVP)

INTERVENTIONS:
Drug: Zidovudine (AZT)+ Didanosine (ddI)+ Nevirapine (NVP) — Zidovudine (AZT) 300mg bid Didanosine (ddI) 200mg bid (W>60Kg)125mg bid (W<60Kg) Nevirapine (NVP) 200mg bid
  Arms: A
Drug: Stavudine (d4T), Lamivudine (3TC), Nevirapine (NVP) — Stavudine (d4T) 30mg bid (W>60Kg)20mg bid (W<60Kg) Lamivudine (3TC)300mg qd Nevirapine (NVP)200mg bid
  Arms: B
Drug: Zidovudine (AZT), Lamivudine (3TC), Nevirapine (NVP) — Zidovudine (AZT) 300mg bid Lamivudine (3TC) 300mg qd Nevirapine (NVP) 200mg bid
  Arms: C

SUMMARY:
The purpose of this study is to determine whether the three generic nevirapine-based antiretroviral regimens are effective in the treatment of Acquired immune deficiency syndrome .

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* the subjects were HIV-seropositive by standard serum enzyme-linked immunosorbent assay (ELISA) tests and also by Western blot analysis
* the subjects were antiretroviral drug-naïve
* a baseline CD4+ T-cell count from 100 to 350 cells/mm3 and a baseline plasma viral load over 500copies/ml

Exclusion Criteria:

* pregnancy or breastfeeding
* anticipated nonadherence
* AIDS-defining illness within 2 weeks of entry
* white blood cell count less than 2.0×109/L, absolute neutrophil count less than 1.0×109/L, hemoglobin level less than 90g/l, platelet count less than 0.75×1012/L
* transaminase and alkaline phosphatase level more than 3 times the upper limit of the normal range, bilirubin level more than 2.5times the upper limit of the normal range, serum creatinine level more than 1.5 times the upper limit of the normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2005-01; Primary Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Li T, Dai Y, Kuang J, Jiang J, Han Y, Qiu Z, Xie J, Zuo L, Li Y. Three generic nevirapine-based antiretroviral treatments in Chinese HIV/AIDS patients: multicentric observation cohort. PLoS One. 2008;3(12):e3918. doi: 10.1371/journal.pone.0003918. Epub 2008 Dec 12. PMID 19081791